CLINICAL TRIAL: NCT05477615
Title: Phase II Trial of Lazertinib and Pemetrexed/Carboplatin Combination in Patients With EGFR Positive, Metastatic NSCLC With Asymptomatic or Mild Symptomatic Brain Metastases After Failure of Osimertinib
Brief Title: Lazertinib/Pemetrexed/Carboplatin After Osimertinib Failure in NSCLC With Brain Metastases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jin Hyoung Kang (Other)
Collaborators: Korea University Anam Hospital (Other)
Responsible Party: Sponsor-Investigator, Jin Hyoung Kang, Professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LU21-17
Record Dates: First submitted 2022-07-17; First posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — lazertinib; Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- lazertinib/pemetrexed/carboplatin (Experimental): combination of lazertinib with pemetrexed/carboplatin chemotherapy
  - Lazertinib 240mg once daily and chemotherapy (pemetrexed and carboplatin) is administered on the 1st day every 3 weeks.
  Interventions: Drug: Lazertinib; Drug: Pemetrexed; Drug: Carboplatin

INTERVENTIONS:
Drug: Lazertinib — - Lazertinib 240mg (3 tablets, 80mg/1tablet) once a day, oral, before disease progression
  Other Names: YH25448
Drug: Pemetrexed — - Pemetrexed 500mg/m2 is administered on the 1st day every 3 weeks. One cycle of treatment is defined as continuous administration for 21 days. Pemetrexed and carboplatin can be administered in reduced doses according to the principles of each institution.
Drug: Carboplatin — - Carboplatin AUC x 5 mg/mL.min is administered on the 1st day every 3 weeks. One cycle of treatment is defined as continuous administration for 21 days. Pemetrexed and carboplatin can be administered in reduced doses according to the principles of each institution.

SUMMARY:
The primary objective is to evaluate the intracranial efficacy of pemetrexed/carboplatin chemotherapy and lazertinib combination therapy after osimertinib failure in EGFR-positive non-small cell lung cancer patients with brain metastasis. The primary endpoint is the incracranial objective response rate (iORR). Secondary endpoints are intracranial progression free survival, (iPFS), objective response rate (ORR), duration of response (DoR), disease control rate, (DCR), overall survival (OS), the pattern of treatment failure, intracranial salvage treatment rate, and toxicity.

Patients should take lazertinib 240 mg (80 mg, 3 tablets) once a day at the same time as possible before meals. Chemotherapy will be administered on the 1st day every 3 weeks. (Pemetrexed 500mg/m2, Carboplatin AUC x 5 mg/mL.min) One cycle of treatment is defined as continuous administration for 21 days.

The treatment will be applied to the all patients until documented evidence of disease progression, unacceptable toxicity, noncompliance, or withdrawal of consent, or the investigator decides to discontinue treatment, whichever comes first. If the investigator decides to reduce the dose due to an adverse reaction during the administration of lazertinib 240 mg, the dose may be reduced to 160 mg (80 mg, 2 tablets) of lazertinib. Pemetrexed and carboplatin can be administered in reduced doses according to the principles of each institution.

DETAILED DESCRIPTION:
The primary objective is to evaluate the intracranial efficacy of pemetrexed/carboplatin chemotherapy and lazertinib combination therapy after osimertinib failure in EGFR-positive non-small cell lung cancer patients with brain metastasis. The primary endpoint is the incracranial objective response rate (iORR), defined as the proportion of patients achieving a complete response or partial response of intracranial lesions per RECIST v1.1 by investigator's assessments. Secondary endpoints are intracranial progression free survival, (iPFS), objective response rate (ORR), duration of response (DoR), disease control rate, (DCR), overall survival (OS), the pattern of treatment failure, intracranial salvage treatment rate, and toxicity.

Intracranial objective response rate (iORR): percentage of subjects with at least one confirmed response (CR or PR or responding) in the intracranial lesion before evidence of progression in patients with brain metastases Intracranial progression free survival (iPFS): From C1D1 to the date of either disease progression of intracranial lesions or death Objective response rate (ORR): proportion of patients achieving a complete response or partial response of overall lesions Duration of response (DoR): From the first recorded response to the first recorded disease progression or death Disease control rate, (DCR): proportion of patients achieving a complete response or partial response or stable disease of overall lesions Overall survival: From C1D1 to the date of all-cause mortality Safety: Evaluated by NCI-CTCAE v5.0 Pattern of treatment failure: intracranial progression, extracranial progression, or both Intracranial salvage treatment rate: Percentage of subjects who underwent salvage treatment(surgery or radiation) due to intracranial disease progression

The exploratory objective is to identify molecular profiling using next generation sequencing.

Patients should take lazertinib 240 mg (80 mg, 3 tablets) once a day at the same time as possible before meals. Chemotherapy will be administered on the 1st day every 3 weeks. (Pemetrexed 500mg/m2, Carboplatin AUC x 5 mg/mL.min) One cycle of treatment is defined as continuous administration for 21 days.

The treatment will be applied to the all patients until documented evidence of disease progression, unacceptable toxicity, noncompliance, or withdrawal of consent, or the investigator decides to discontinue treatment, whichever comes first. If the investigator decides to reduce the dose due to an adverse reaction during the administration of lazertinib 240 mg, the dose may be reduced to 160 mg (80 mg, 2 tablets) of lazertinib. Pemetrexed and carboplatin can be administered in reduced doses according to the principles of each institution. To prevent side effects of pemetrexed, start at least 7 days before cycle 1 daily dose of 350-1,000 μg/day of folic acid and 1000 μg/3 of vitamin B12.

ELIGIBILITY:
Inclusion Criteria:

1. Written consent A. Patients who voluntarily provided written informed consent prior to participation in the clinical trial B. Patients who voluntarily provide written informed consent for genetics and/or exploratory studies
2. Age and gender A. Male or female, 20 years of age or older B. Female patients must agree to the use of appropriate contraceptive methods and not be lactating, and for women of childbearing age, there must be evidence that the pregnancy test is negative prior to initiation of dosing, or that they are not fertile because they meet one of the following criteria at screening: box "Postmenopausal" women over the age of 50 and who are amenorrhea for at least 12 months after stopping all exogenous hormone therapy Records of irreversible surgical infertility by hysterectomy, bilateral ovariectomy, or bilateral yolk resection, tubal ligation are not permitted Women under 50 years of age had amenorrhea for at least 12 months after stopping all exogenous hormone therapy, and the levels of luteinizing hormone (LH) and follicle stimulating hormone (FSH) were within the postmenopausal range of the laboratory. Is only recognized as a postmenopausal condition C. Male patients who have not undergone vasectomy must consent to the use of a blocking contraception method, i.e., condom, and sperm supply is prohibited until 3 months after taking the last investigational drug D. Must be able to swallow tablets
3. Target disease A. Histologically or cytologically confirmed locally advanced or metastatic non-small cell lung cancer patients. This may occur as systemic recurrence after prior surgery for early stage disease or patients may be newly diagnosed with stage IIIB/C or IV disease.

B. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-2, with no deterioration in the last 2 weeks C. Life expectancy judged by the Investigator of at least 3 months D. Disease status

* Confirmed sensitizing EGFR mutation prior to administration of osimertinib (L858R, Exon 19 deletion, G719X and L861Q mutations should be confirmed as a record)
* Failure after osimertinib. Past treatment history for locally advanced or metastatic NSCLC limited to two regimen of EGFR TKI treatment (osimertinib and/or gefitinib, erlotinib, or afatinib) and/or one palliative cytotoxic chemotherapy regimen (A wash-out period of at least 2 months is required until administration after the last dose of osimertinib)
* Asymptomatic or mild symptomatic brain metastases progressed or newly confirmed patients
* One or more intracranial measurable disease in accordance with Response Evaluation Criteria in Solid Tumors (RECIST v 1.1). The target lesion that has received previous local therapy should not be considered as measurable. However, new CNS lesion after more than 3 months of previous local therapy could be considered as target lesion.

Exclusion Criteria:

* 1) The following interventional treatment A. Prior treatment with lazertinib B. Prior treatment with investigational drugs in other clinical trials within 30 days prior to the first administration C. Patients who received cytotoxic chemotherapy for the treatment of advanced non-small cell lung cancer or other anticancer drugs other than EGFR TKI within 14 days prior to the first administration of the investigational drug D. Prior local-regional therapy within 4 weeks prior to Day 1 of trial treatment (e.g., major surgery, radiation therapy [with the exception of palliative bone-directed radiotherapy and radiotherapy administered to superficial lesions], hepatic arterial embolization, transcatheter arterial chemoembolization, chemoembolization, radiofrequency ablation, percutaneous ethanol injection, or cryoablation) G. Patients currently receiving drugs or herbal supplements known as inhibitors or inducers of CYP3A4 or who cannot discontinue use at least 1 week prior to the first dose of lazertinib.

H. Previous anticancer treatment-related toxicities not recovered to baseline or Grade 0-1 (except alopecia) 2) Medical history and current disease A. Symptomatic spinal cord compression (However, registration is allowed if steroid treatment is not required within at least 2 weeks before the start of administration of the investigational drug) B. Symptomatic and unstable central nervous system (CNS) or brain metastasis requiring local treatment at screening. (Asymptomatic or mild symptomatic leptomeningeal metastasis is also permitted to be registered) C. Symptomatic or intracranial bleeding that needs treatment D. History of interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD E. Carcinoma other than non-small cell lung cancer, if the investigator is judged to be inadequate to participate in this clinical trial due to evidence of severe or uncontrolled systemic disease, uncontrolled hypertension, or active bleeding tendency, or that it is difficult to follow this protocol. (Screening for chronic disease is not required)

F. Any of the following cardiovascular diaseases:

i. A history of congestive heart failure (CHF) of grade 3 or higher according to the New York Heart Association Classification (NYHA) or cardiac arrhythmia requiring treatment ii. A History of unstable angina or myocardial infarction experienced within 6 months before the first administration of the investigational drug iii. Left ventricular ejection fraction <45% on recent echocardiography or MUGA scan G. Known human immunodeficiency virus (HIV) infection H. Patients with refractory nausea and vomiting, chronic gastrointestinal disorders, inability to swallow the product, or undergoing enterectomy deemed to interfere with the proper absorption of lazertinib.

I. History of hypersensitivity to drugs J. Clinically significant chronic infection or major medical or mental illness K. Subjects with any concurrent medical condition or disease that will potentially compromise the conduct of the study at the discretion of the Investigators L. History of allogeneic hematopoietic stem cell transplantation, history of whole blood transfusions that did not remove leukocytes within 120 days before the date of collection of genetics specimens 3) Criteria for cardiology and clinical laboratory testing

A. Cardiac criteria in any of the following:

i. Based on the QTc value measured with an electrocardiogram (ECG) device during screening, the average of the correction of the QT interval (QTc) at rest on an electrocardiogram (ECG) measured three times> 470 msec ii. Clinically important abnormalities of rhythm, conduction, or shape on the ECG at rest. For example, complete left block, 3rd degree cardiac block, 2nd degree cardiac block, PR interval> 250 msec iii. Increased risk of QTc prolongation or arrhythmia, such as heart failure, hypokalemia, congenital QT prolongation syndrome, concomitant medications known to prolong QT intervals, QT prolongation syndrome or a family history of unexplained sudden deaths under 40.

B. Laboratory index at baseline:

iv. Hemoglobin ≤ 8.0 g/dL (without transfusion or growth factor support in the preceding 14 days) v. Neutrophils < 1.0 x 109/L vi. Platelets < 100 x 109/L (without transfusion or growth factor support in the preceding 7 days) vii. Total bilirubin > 3 mg/dL viii. Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) > 5 x upper limit of normal (ULN) ix. Renal impairment as evidenced by serum creatinine ≥ 1.5 x ULN, or calculated creatinine clearance (CrCl) < 50 mL/min by Cockroft-Gault formula (24-hour CrCl might be requested by the Investigator for confirmation, if calculated CrCl is < 60 mL/min. In such case, subjects with 24-hour CrCl < 50 mL/min should be excluded)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
intracranial objective response rate | "every 6 weeks up to 24 weeks, and every 12 weeks thereafter up to 2 years "
  "Percentage of subjects who had at least one confirmed response among evaluable subjects who performed more than one response assessment"

SECONDARY OUTCOMES:
intracranial progression-free survival | "every 6 weeks up to 24 weeks, and every 12 weeks thereafter up to 2 years "
  "The period (in months) from the first administration of the investigational drug to the date of onset of objective intracranial disease progression evaluated by the investigator or death from any cause, whichever occurs first"
overall response rate | every 6 weeks up to 2 years
  the percentage of subjects who had at least one complete response (CR) or partial response (PR) with a confirmed response (RECIST 1.1) before evidence of disease progression appeared
duration of response | every 6 weeks up to 2 years
  the time from the first documented date of a later confirmed response to the date of documented disease progression or death (equivalent to the occurrence of the PFS event), whichever occurs first.
disease control rate | every 6 weeks up to 2 years
  the percentage of subjects with a Best Overall Response (BOR), extracranial and intracranial response of CR, PR, responding, or SD.
overall survival | every 6 weeks up to 2 years
  the period from the first administration of the investigational drug to the date of death of any cause.
pattern of treatment failure | every 6 weeks up to 2 years
  intracranial disease progression or extracranial disease progression, or both
salvage intracranial treatment rate | every visit up to 2 years
  the percentage of subjects who received salvage treatment (brain radiation or surgery) due to intracranial disease progression.
adverse events | every visit up to 2 years
  All subjects receiving at least one dose of Lazertinib will be included in the safety profile evaluation (safety analysis cohort).

CONTACTS AND LOCATIONS:
Overall Officials: Jin Hyoung Kang, Study Chair — Seoul St. Mary's Hospital, The Catholic University of Korea
Locations (6):
- South Korea (6):
  - Gachon University Gil Medical Center, Gyeonggi-do
  - Incheon St. Mary's hospital, Catholic university of Korea, Incheon
  - Gachon University Gil Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hosptial, Seoul
  - Seoul St. Mary's Hospital, Catholic University of Korea, Seoul

IPD SHARING:
Plan to Share IPD: No